CLINICAL TRIAL: NCT06163443
Title: Evaluating the Impact of B Vitamin Supplementation (Soloways™) on Homocysteine and LDL-C Levels in Patients With MTHFR, MTR, and MTRR Polymorphisms: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Evaluating the Impact of B Vitamin Supplementation (Soloways™) on Homocysteine and LDL-C Levels in Patients With MTHFR, MTR, and MTRR Polymorphisms.
Acronym: VITAGEN-H
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Triangel Scientific (Industry); Center of New Medical Technologies (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SW002
Record Dates: First submitted 2023-11-22; First posted 2023-12-08 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hyperhomocysteinemia; Hyperlipoproteinemias
Keywords: Methylfolate; Homocysteine; Genetic Polymorphisms (MTHFR, MTR, MTRR); Cardiovascular Risk; Methylcobalamin; LDL-C; Cholesterol; Low-Density Lipoprotein
MeSH Terms: conditions — Hyperhomocysteinemia; Hyperlipoproteinemias | interventions — Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin B group (Experimental): Patients with polymorphisms in the MTHFR, MTR, and MTRR will take methylfolate, P5P, and methylcobalamin genes 2 capsules/day.
  Interventions: Dietary Supplement: Vitamin B
- Placebo group (Placebo Comparator): Patients with polymorphisms in the MTHFR, MTR, and MTRR will take placebo capsules will be identical in appearance, matched for color coating, shape, and size - 2 capsules/day..
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin B — MTHFR, MTR, and MTRR polymorphysm based L-methylfolate (1 mg), P5P (pyridoxal-5-phosphate, 50 mg), and Methylcobalamin (500 mcg) prescription
  Arms: Vitamin B group
Dietary Supplement: Placebo — MTHFR, MTR, and MTRR polymorphysm based placebo prescription
  Arms: Placebo group

SUMMARY:
This randomized, double-blind, placebo-controlled trial will evaluate the impact of methylfolate, pyridoxal-5'-phosphate (P5P), and methylcobalamin supplementation on homocysteine and LDL-C levels in individuals with low to medium cardiac risk and MTHFR, MTR, and MTRR gene polymorphisms. The study aims to explore the efficacy of these vitamins in reducing homocysteine levels, a critical risk factor for cardiovascular disease (CVD), while also monitoring LDL-C levels. The findings will offer valuable insights into personalized CVD prevention and management, emphasizing the significance of genetic factors in nutritional therapy.

DETAILED DESCRIPTION:
Design: Participants with specific genetic polymorphisms and homocysteine levels above 15 µmol/L, without a history of severe CVD or other exclusion criteria, will be enrolled and randomized into two groups: one receiving methylfolate, P5P, and methylcobalamin, and the other a placebo. The study, adhering to ethical standards and informed consent, will involve 54 patients divided equally between the treatment and placebo groups. The primary endpoint will be the percent change in homocysteine levels over six months, with secondary endpoints including changes in LDL-C and other lipid profile components.

Intervention: Participants will receive either the active treatment (L-methylfolate, P5P, and Methylcobalamin) or a placebo, with both groups taking two capsules daily for 180 days. Fasting measurements of lipid profiles and homocysteine levels will be conducted at the start, midpoint, and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75.
* Homocysteine levels greater than 15 µmol/L and LDL-C level between 70 and 190 mg/dL, confirmed in at least two sequential checks conducted within the last six months prior to signing the consent form.
* Presence of at least one minor allele in any of the following genetic polymorphisms: rs1801133 (MTHFR C677T), rs1801131 (MTHFR A1298C), rs1805087 (MTR A2756G), and rs1801394 (MTRR A66G).

Exclusion Criteria:

* Personal history of cardiovascular disease or high risk (≥ 20%).
* Triglycerides (TG) ≥ 400 mg/dL.
* Obesity (Body Mass Index > 32 kg/m^2).
* Assumption of lipid-lowering drugs or supplements affecting lipid metabolism within the last three months.
* Use of medications or supplements known to affect homocysteine levels, such as B-vitamins and certain antihypertensives, within the last three months.
* Diabetes mellitus.
* Known severe or uncontrolled thyroid, liver, renal, or muscle diseases.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Homocysteine levels | 180 days
  The primary endpoint is the percent change in homocysteine levels from baseline to 6 months of observation, comparing a combined treatment regimen of methylfolate, P5P, and methylcobalamin in MTHFR, MTR, and MTRR polymorphysm.

SECONDARY OUTCOMES:
Change in LDL-C Levels | 180 days
  Percent change in Low-Density Lipoprotein Cholesterol (LDL-C) levels.
Change in HDL-C Levels | 180 days
  Percent change in High-Density Lipoprotein Cholesterol (HDL-C) levels.
Change in Total Cholesterol | 180 days
  Percent change in total cholesterol levels in the study participants.
Change in Serum Triglycerides | 180 days
  Percent change in serum triglycerides.
Change in hsCRP Levels | 180 days
  Percent change in high-sensitivity C-Reactive Protein (hsCRP) levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Center of New Medical Technologies, Novosibirsk, Novosibirsk Oblast, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pokushalov E, Ponomarenko A, Bayramova S, Garcia C, Pak I, Shrainer E, Ermolaeva M, Kudlay D, Johnson M, Miller R. Effect of Methylfolate, Pyridoxal-5'-Phosphate, and Methylcobalamin (SolowaysTM) Supplementation on Homocysteine and Low-Density Lipoprotein Cholesterol Levels in Patients with Methylenetetrahydrofolate Reductase, Methionine Synthase, and Methionine Synthase Reductase Polymorphisms: A Randomized Controlled Trial. Nutrients. 2024 May 21;16(11):1550. doi: 10.3390/nu16111550. PMID 38892484
- See also: 10.3390/nu16111550 — https://pubmed.ncbi.nlm.nih.gov/38892484/